CLINICAL TRIAL: NCT02867865
Title: Perioperative Therapy Preoperative Chemotherapy Versus Chemoradiotherapy in Locally Advanced Gall Bladder Cancers
Acronym: POLCAGB
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Reena Engineer, Professor and Radiation oncologist, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1652
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Gall Bladder Cancers
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Gemcitabine; Cisplatin; Chemoradiotherapy; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy arm (Active Comparator): Post staging laparoscopy, all patients will receive chemotherapy using Injection Gemcitabine 1000 mg/m2 delivered day 1 and 8 every 3 weeks.
  In addition, Injection Cisplatin 25 mg/m2 for and 4 cycles week 1 to week 11.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Procedure: PETCECT; Procedure: Laparoscopy
- Chemoradiation arm (Experimental): Post staging laparoscopy in Experimental arm The radiation dose will be 50-55 Gy/ 25 fractions to the gross disease and 45 Gy/ 25 fractions to suspected microscopic disease along with weekly gemcitabine (300 mg/ m2). Radiotherapy will be for 5 weeks which will be followed by 2 cycles of chemotherapy with Injection Gemcitabine (Gemcite,Gemzar) 1000 mg/m2 delivered day 1 and 8 every 3 weeks and cisplatin (Cisplat, Cytoplatin) 25 mg/m2from week 7 to week 11.
  During week 12-13 patients will undergo repeat PETCECT scan. If the scan shows partial or good response then patients will be evaluated for surgery. Surgery if possible will be done between weeks 13-15. In case of inoperable disease patients will receive further chemotherapy
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: Chemoradiation; Procedure: PETCECT; Procedure: Laparoscopy

INTERVENTIONS:
Drug: Gemcitabine — Those randomized to systemic chemotherapy alone will proceed to receive Chemotherapy Gemcitabine gemcitabine 1000 mg/m2delivered day 1 and 8 every 3 weeks for 4 cycles
  Other Names: Gemcite; Gemzar
Drug: Cisplatin — Inj. cisplatin 25 mg/m2 delivered. day 1 and 8 every 3 weeks for 4 cycles
  Other Names: Cytoplat
Radiation: Chemoradiation — Radiotherapy will be for 5 weeks and will be given only in the study arm. The radiation dose will be 50-55 Gy/ 25 fractions to the gross disease and 45 Gy/ 25 fractions to suspected microscopic disease along with weekly gemcitabine (300 mg/ m2).
  Other Names: Intensity modulated radiotherapy
  Arms: Chemoradiation arm
Procedure: PETCECT — All the patients will undergo PETCECT to rule out metastatic disease
  Other Names: PET scan
Procedure: Laparoscopy — Patients will be subjected to staging laparoscopy with 16b1 lymph node biopsy to rule out metastatic disease.
  Other Names: Diagnostic laparoscopy

SUMMARY:
Locally advanced Gall bladders cancers not amenable for curative resection are often treated with chemotherapy alone which is the current standard of care. Randomized trials have shown survival benefit with combination chemotherapy in gallbladder cancers. Gallbladder cancer is not common western world and thus there is lack of evidence regarding the impact of neoadjuvant or concurrent chemo-radiation in this cancer.Use of neoadjuvant treatment with chemotherapy alone or chemoradiotherapy has shown to downsize these tumors to safely undergo R0 resection in few published studies. Also if the patients develop distant metastasis during this neoadjuvant therapy they can be spared of unnecessary surgery.

In a pilot study of 28 patients by Engineer et al conducted at Tata Memorial centre treated with neoadjuvant concurrent chemoradiation the investigators could achieve R0 resectability rate 0f 47% with a median overall survival (OAS) and progression free survival (PFS) of 35 and 20 months for the patients undergoing R0 resection.

In this study the investigators intend to compare the effects of using neoadjuvant chemotherapy alone vs. neoadjuvant chemoradiation and chemotherapy for locally advanced gall bladder cancers in terms of down staging and overall survival.

DETAILED DESCRIPTION:
Introduction:

Adenocarcinoma of the gallbladder (GBCA) is the most common malignancy of the biliary tract and its incidence is alarmingly high in the Indian subcontinent. Complete surgical excision is the standard of care for both gallbladder and pancreatic cancers. Unfortunately, majority of these cancers are diagnosed at an advanced, inoperable stage and only 10-30% of the patient present with resectable disease.

Gall bladder cancers which are T3/T4 with liver infiltration, with or without visceral/vascular infiltration or having large local lymph node metastases; in the absence of distant metastases are generally considered as locally advanced. There prognosis in terms of resectability and survival remains dismal in most of the reports.

Even with aggressive surgery like extrahepatic bile duct resection or pancreaticoduodenectomy the 5 year survival rate for stage III disease ranges 30% to 42% in best of the reports. But these results are often not reproducible.

Locally advanced Gall bladders cancers not amenable for curative resection are often treated with chemotherapy alone which is the current standard of care. Randomized trials have shown survival benefit with combination chemotherapy in gallbladder cancers. In a randomized trial combination chemotherapy of Gemcitabine and cisplatin was superior to Gemcitabine chemotherapy alone and local tumor response in terms of partial downsizing or stable disease was achieved in 81% of cases. With Gemcitabine and Cisplatin based Neoadjuvant chemotherapy (NACT) some locally advanced GB cancers do get downstaged to undergo resection. Recent publication from Tata Memorial Centre, where NACT alone was given which resulted in surgical resection rate of 43% median OAS and PFS being 13 months and 8 months.

Study methodology:

All patients with diagnosis of non metastatic locally advanced Gall bladder cancers who fulfill the study eligibility criteria will be evaluated for study participation and will undergo Positron emission tomography and contrast enhanced computerized tomography (PETCECT) scan and staging laparoscopy to rule out metastatic disease. Patients will undergo upfront randomization into one of the study arms.

A proportion of patients are expected to have jaundice or cholangitis at presentation. At study inclusion there should be no clinical evidence of active cholangitis or unresolved biliary obstruction. Liver Function Tests, Renal Function Tests and CA 19-9 within 4 weeks of treatment initiation.

Systemic Chemotherapy arm (Standard Arm or Arm A)

Those randomized to NACT will proceed to receive systemic gemcitabine 1000 mg/m2delivered day 1 and 8 every 3 weeks and cisplatin 25 mg/m2 for and 4 cycles (week 1- week 11).

Chemoradiation arm (Study Arm or Arm B)

The radiation dose will be 50-55 Gy/ 25 fractions to the gross disease and 45 Gy/ 25 fractions to suspected microscopic disease along with weekly gemcitabine (300 mg/ m2). Radiotherapy will be for 5 weeks which will be followed by 2 cycles of chemotherapy (week 7 to week 11)

These radiotherapy (RT) doses have found to be safe in the investigators pilot study.

During week 12-13 patients will undergo repeat PETCECT scan. If the scan shows partial or good response then patients will be evaluated for surgery. Surgery if possible will be done between weeks 13-15. In case of inoperable disease patients will receive further chemotherapy. With locally progressive/systemic disease on chemotherapy patients may be considered for second line palliative chemotherapy or best supportive care. The use of radical dose chemoradiation is not allowed on disease progression in the systemic chemotherapy arm. However palliative radiation may be used.

Surgery

Surgical procedure will be en-bloc resection including cholecystectomy with a liver wedge excision and periportal lymph node clearance. Nodal clearance from station number 8, 12, 13 with sampling of inter aortocaval node will be done. Extrahepatic biliary excision or additional organ excision will be done as per the discretion of operating surgeon.

Post Surgery all patients will receive additional adjuvant chemotherapy

Number of patients enrolled: Screened 350 Enrolled 314

ELIGIBILITY:
Inclusion Criteria:

Locally advanced T3 or T4 tumors with one or more of the following:

-> 2 cm but < 5 cm liver invasion

* Radiological involvement of antropyloric region of stomach, duodenum, hepatic flexure of colon or small intestine, but without infiltration of the mucosa on endoscopy.
* Type I/II invasion -Involvement of bile duct (common hepatic duct or proximal 1/3 of the common bile duct) causing obstructive jaundice
* Radiological suspicion of lymph node involvement N1 {stations 8, 12, 13) Hepatic artery (Station 8), hepatoduodenal ligament (Station 12), retropancreatic/retroduodenal (Station 13) i.e. size>1cm in short axis, round in shape, and heterogenous enhancement on PET scan.
* Vascular involvement : impingement/ involvement (<180 degree angle) of one or more of the following blood vessels common hepatic artery/ right hepatic artery/main portal vein/right portal vein (stage III disease)
* Patient who have undergone prior cholecystectomy having residual disease with at least one of the above features.
* Biopsy/ cytology proven adenocarcinoma
* More than 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 Normal hematological and renal and hepatic functions (serum bilirubin < 3mg/dl)

Exclusion Criteria:

* Resectable disease
* Evidence of distant metastasis (Liver, Lung, peritoneum, port site etc)
* Involving major part of the liver precluding restriction of full RT doses
* Received any prior radiation or chemotherapy.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 6 years
  To compare the Overall survival between the patients treated with neoadjuvant chemotherapy alone vs. patients treated with neoadjuvant chemoradiation. Overall survival will be calculated from the date of randomization to the date of death

SECONDARY OUTCOMES:
Surgical resection rate | 6 years
  R0 surgical resection rate would be compared in patients who undergo complete resection.
Progression free survival | 6 years
  Progression free survival between the two groups. survival will be calculated from the date of randomization to the date of progression whether local or distal.
Number of participants with treatment related serious adverse events | From the start of treatment until 30 days after the end of treatment, up to approximately 14 months
  Adverse events are assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Adverse events are considered to be related to treatment if the Investigator deems them to be either possibly, probably, or definitely related to treatment Acute toxicities will be measured within 12 weeks of completeion of neoadjuvant Radiotherapy or Chemotherapy
Deterioration free rate of quality of life (QOL) scores at baseline and three monthly | Upto 2 years
  QOL questionnaires will be applied to patients at baseline and every 12 weeks for a maximum of 12 months. The secondary endpoint will be analysed at the end of the study. FACT (Functional Assessment of Cancer Therapy) -Hep (Hepatic) version 4 will be used to assess quality of life for all patients. It will be assessed at baseline then at the completion of neoadjuvant treatment thereafter 3 monthly at every follow up

CONTACTS AND LOCATIONS:
Overall Officials: Reena Engineer, MBBS MD, Principal Investigator — Professor and Radiation oncologist
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Engineer R, Patkar S, Lewis SC, Sharma AD, Shetty N, Ostwal V, Ramaswamy A, Chopra S, Agrawal A, Patil P, Mehta S, Goel M. A phase III randomised clinical trial of perioperative therapy (neoadjuvant chemotherapy versus chemoradiotherapy) in locally advanced gallbladder cancers (POLCAGB): study protocol. BMJ Open. 2019 Jun 27;9(6):e028147. doi: 10.1136/bmjopen-2018-028147. PMID 31253621